CLINICAL TRIAL: NCT00901849
Title: Phase 1 Study of Tarceva and Rapamycin For Recurrent Low-Grad Gliomas in Children With or Without Neurofibromatosis Type 1 (NF1)
Brief Title: Tarceva/Rapamycin for Children With Low-grade Gliomas With or Without Neurofibromatosis Type 1 (NF1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roger Packer (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor-Investigator, Roger Packer, Senior Vice President, Center for Neuroscience and Behavioral Medicine;, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4104
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Low-grade Gliomas
MeSH Terms: interventions — Erlotinib Hydrochloride; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tarceva and Rapamycin — Tarceva will be administered once a day for 28 days without interruption. THen Rapamycin will be administered, orally twice daily, in combination with the Tarceva for the remainder of the study.

SUMMARY:
This study will evaluate the feasibility of combining two drugs, Tarceva (an anti-EGFR agent), and Rapamycin (an mTOR inhibitor), in children with progressive low-grade gliomas who have failed initial conventional treatment. In addition to evaluating the toxicity of this drug regimen, the potential efficacy of the regimen will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* children less than 21 years of age, with or without neurofibromatosis, with recurrent low-grade gliomas.
* patients with or without NF1 must have failed some form of conventional therapy, radiotherapy, or chemotherapy (carboplatin/vincristine) to be eligible, including those treated wtih initial surgery. Patients do not have to have received radiotherapy to be eligible.
* children with all types of histologically proven low-grade gliomas will be eligible; re-operation at the time of recurrence is not mandatory for entry on study.
* patients with intrinsic brain lesions, believed neuroradiographically consistent with a low-grade glial tumor, with neurofibromatosis type 1 can be treated without histological confirmation.
* patients without neurofibromatosis type 1 must have histological confirmation of a low-grade glial tumor prior to entry on study.
* patients must have a Karnofsky score of greater than or equal to 50% for children greater than 10 years of age, or a Lansky score of greater than or equal to 50% for patients less than 10 years of age.
* patients who are unable to walk because of paralysis, but who are able to use a wheelchair, will be considered ambulatory for purposes of assessing performance score.
* patients must have a life expectancy of at least 12 weeks.
* patients must be able to swallow medication in tablet form.
* patients must have adequate organ function, including: peripheral ANC of greater than 1,000/microliters; a platelet count of greater than 100,000/microliters; hemoglobin of greater than 8 gms,dl (pRBC transfusions of allowed to maintain hemoglobin > 8 g/dl)
* patients must have adequate renal function, which is defined as a normal serum creatinine for age
* patients must have adequate liver function, as defined as a total bilirubin or less than 1.5 times the upper limit of normal for age, and an SGPT (ALT) of less than 2.5 times the upper limit of normal for age
* patients must have had a MR scan within 3 weeks of starting treatment
* all patients, and/or their parents or legal guardian, must sign a recent informed consent
* all institutional, FDA, and NCI requirements for human study must be met.

Exclusion Criteria:

* patients must not have any other active tumors.
* pregnancy or breast feeding is an exclusion criteria, as the potential mutagenicity and cytotoxicity of these drugs in developing fetuses are unknown. A pregnancy test must be obtained in females who are postmenarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* patients with uncontrolled infection are excluded.
* patients who have previously received Tarceva or Rapamycin are excluded.
* patients on antiepileptics and/or corticosteroids are allowed on study as long as they have been on a stable or weaning dose for 7 days prior to study initiation (defined as first day of treatment).

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Participants will remain on the trial for one year if benefiting from drug as demonstrated by radiographic evaluation and clinical evaluation. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Research Institute, Washington D.C., District of Columbia, United States